CLINICAL TRIAL: NCT04112706
Title: Efficacy of CPP-ACP on Bleaching Related Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New England (Other)
Collaborators: University of Iowa (Other)
Responsible Party: Principal Investigator, Shaista Rashid, Assistant Clinical Professor, University of New England
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB 200604706
Record Dates: First submitted 2019-09-24; First posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Teeth Sensitivity; Tooth Discoloration
MeSH Terms: conditions — Dentin Sensitivity; Tooth Discoloration | interventions — casein phosphopeptide-amorphous calcium phosphate nanocomplex

STUDY DESIGN:
Intervention Model Description: Randomized controlled split-mouth
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: CPP-ACP — CPP-ACP WAS APPLIED AFTER TOOTH BLEACHING

SUMMARY:
Objective: The purpose of this randomized controlled split-mouth clinical trial was to evaluate the effectiveness of MI paste in reducing sensitivity associated vital bleaching.

Methods: 45 subjects were randomly divided into two groups, based upon which arch received MI Paste. Group 1 bleached Maxillary arch, Group 2 bleached mandibular arch. Two weeks later subjects stopped bleaching the first arch and started second arch. Sensitivity was measured by VAS daily log scale for two weeks. Shade was taken with colorimeter and Classic Vita shade guide at baseline, immediate post-bleaching, and two weeks post-bleaching. Longitudinal sensitivity over the 14 days period of bleaching was summarized. The Wilcoxon Signed Rank test was used to compare summary measures.

DETAILED DESCRIPTION:
Study Design

This was a randomized, controlled, split-mouth cross-over design clinical trial. Subjects were randomized into two groups depending on the control and intervention arches:

* Group 1: The maxillary arch was the control arch (only bleaching) while the mandibular arch (MN) was intervention arch (bleaching and MI Paste).
* Group 2: The MN arch was the control arch (only bleaching) while the MX arch was the intervention arch (bleaching and MI Paste).

Ethical permission for the study was obtained from the University Intuitional Review Board (No. 200604706). The study was conducted in full accordance with the Helsinki Declaration and reported using CONSORT guidelines. Informed consents were obtained from the subjects prior to enrolment in the study.

Participants Forty-six participants were recruited at the Oral Health Center. Participants were included if they age between 18 and 55 years old with no prior history of bleaching, not using any desensitizing agents, and with anterior teeth of shade A2 or higher. Participants allergic to milk protein, pregnant, and/or on daily NSAIDs were excluded. They were also excluded if they have had an anterior crown or composite restoration, scaling or periodontal surgery performed in the past six months, and/or had a history of bleaching.

Intervention Both the bleaching gel (TiON whitening gel (GC America Inc) and MI paste (PROSPECTM MI paste) were delivered using custom trays with reservoir made for participants at the beginning of the study. To avoid contamination, the control arch was always bleached first. Group 1 subjects were instructed to use 15% carbamide peroxide on maxillary arch while group 2 were instructed to use it on the mandibular arch. Subjects stopped bleaching on their respective arches after 2 weeks. Subjects were then given bleach and MI paste to be used on the opposing arch (Group 1 used it on the mandibular arch and Group 2 used it on maxillary arch).

For bleaching only arch, participants were instructed to wear the trays each night for 6-8 hours for two weeks. Subjects were given a VAS daily log to document the sensitivity for two weeks. For bleach and MI Paste arch, participants were instructed to brush and floss their teeth, load the non-scalloped tray with MI Paste, wear it for 5 minutes, remove the tray, spit out the excess, and not to eat or drink for one hour. They were instructed to bleach after that for 6-8 hours for the next two weeks. Participants were instructed not to bleach the first arch anymore. Participants were given a VAS daily log to document the sensitivity score for each day for two weeks.

Measurements Measurements were made at baseline (Time 0), 2 weeks after initiation of bleaching (Time 1) and 2 weeks after the end of treatment (i.e., 4 weeks after initiation of bleaching; Time 2) for each arch. Longitudinal VAS scores were to be assessed at baseline (Day 0) and daily during the two weeks of bleaching (Days 1 through 14).

Sensitivity Sensitivity was measured using thermal sensitivity scale (VAS) of 0-10, with 0 being "no pain" and 10 being "severe pain." Subjects were asked to pick a number. Thermal sensitivity was measured by using a 1-second air blast at 70oF from dental unit air syringe as per American Dental Association (ADA) guidelines. A Scale of 0-3 was used to measure the pain response with 0 indicating "no pain" and 3 indicating the "severe pain" which lasted for more than 10 seconds12.

Shade Value-oriented Vita classical shade guide was used to determine the shade of the teeth under standardized conditions for color corrected light. Shade scores were ordered from 1 to 16 according to the brightness grouping recommended by the manufactures. A hand held coloriometer "Shade Vision" (X-rite, Inc) was used to measure shade digitally. Shade Vision identifies color difference using three dimensional CIE L*a*b* values system.

Participants' Survey Participants were given a survey at the end of the study examining their perception on the ease of application of MI Paste as well as the impact of MI Paste on sensitivity and gingival inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between the age of 18 and 50 years who were capable of providing informed consent. Subjects older than 50 were not included in the study because of more secondary dentine present less chances of developing sensitivity.
* Subject who had anterior tooth discoloration (equivalent to or darker than Vita shade A3).
* Subjects who were available for a potential recall period of one year.
* Subjects who had no severe systemic disorders. Subjects who needed antibiotics for prevention of spontaneous bacterial endocarditis (SBE) or artificial joints were included.

Exclusion Criteria:

* Subjects who had any known allergies to any materials used in this protocol.
* Patients with milk protein allergies since one of the materials used is derived from milk protein.
* Pregnant women were excluded from the study due to lack of available data for the safety of the bleaching gel for pregnant women.
* Subjects involved in other clinical trials utilizing a similar protocol.
* Subject who had used any dentist-supplied or over the counter vital tooth bleaching product in the previous six months.
* The subjects who have used any desensitizing agents including toothpaste in the past six months.
* Subjects who took COX-2 NSAIDs on daily basis or were under medical treatment at that time for major psychiatric illness that may have altered the perception of pain/discomfort and/or inhibit the subject from completing the study.
* Subjects who had any periodontal surgery or scaling performed in the past six months.

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2006-07-16 (Actual); Primary Completion 2007-02-16 (Actual); Study Completion 2007-03-16

PRIMARY OUTCOMES:
Change in sensitivity measures related to bleaching: Subjective Sensitivity | 28 DAYS
  Thermal Sensitivity: Subjective Measure:
  Sensitivity was measured using thermal sensitivity scale (VAS) of 0-10, with 0 being "no pain" and 10 being "severe pain". Subjects were asked to pick a number.
  2. Objective Measure: Thermal sensitivity was measured by using a 1-second air blast at 700F from dental unit air syringe as per American Dental Association (ADA) guidelines. A Scale of 0-3 was used to measure the pain response with 0 indicating "no pain" and 3 indicating the "severe pain" which lasted for more than 10 seconds.
Change in sensitivity measures related to bleaching: Objective Sensitivity | 28 days
  Objective Measure:
  Thermal sensitivity was measured by using a 1-second air blast at 700F from dental unit air syringe as per American Dental Association (ADA) guidelines. A Scale of 0-3 was used to measure the pain response with 0 indicating "no pain" and 3 indicating the "severe pain" which lasted for more than 10 seconds.

SECONDARY OUTCOMES:
Shade change and interference of CPP-ACP with bleaching | 14 days
  Shade:
  1. Subjective shade measurement: Value oriented Vita classical shade guide was used to determine the shade of the teeth under standardized conditions for color corrected light. Shade scores were ordered from 1 to 16 according to the brightness grouping recommended by the manufactures.
  2: Objective shade measurement: "Shade vision" (X-rite, inc) was used to take digital color images with colorimetric filtering technology.

CONTACTS AND LOCATIONS:
Locations (1):
- University of New England, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No